CLINICAL TRIAL: NCT01685463
Title: Transcranial Magnetic Stimulation Used to Both Measure Cortical Excitability and Explore Methamphetamine Cue Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIH/NIDA P20 DA022658; P20DA022658 (NIH)
Record Dates: First submitted 2012-09-10; First posted 2012-09-14 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine, craving, TMS, cortical excitability, prefrontal cortex
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): Transcranial magnetic stimulation (TMS) is a noninvasive brain stimulation technology that can focally stimulate the brain of an awake individual. The brain stimulation techniques could theoretically improve the efficacy of smoking cessation.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Placebo Comparator): Sham-TMS procedures: After rTMS determination, participants were fitted with two electrodes on the scalp just below the hairline. Electrodes will be connected to an Epix VT Transcutaneous Electrical nerve stimulation device.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Active TMS:1 Hz, 100% motor threshold TMS for 15 minutes, total 900 pulses. Electrical stimulation instead.
  Other Names: Magstim Rapid
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — The electrical current of the sham system is titrated to a level matching participants' ratings of active TMS. The sham-TMS scalp discomfort will be matched to that of active TMS.
  Other Names: Epix VT Transcutaneous Electrical Nerve Stimulation Device
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
Specific Primary Aims include:

Aim # 1. The investigators explore the feasibility of using the TMS to investigate the cortical excitability and to inhibit meth cue craving in meth dependent population. The investigators anticipate that meth elevates cortical excitability measured by motor threshold, causes changes of cortical silent period, and RC. The investigators also anticipate that paired pulse measures (short-interval intracortical inhibition, short-interval intracortical facilitation and long-interval intracortical inhibition) will be different from healthy control, which are more directly linked to glutamatergic cortical facilitation and GABAergic inhibition, respectively.

Aim # 2. Given the change of the cortical excitability in meth users, the investigators will use inhibiting TMS (1 Hz) over medial prefrontal cortex to study whether TMS can be used to reduce cue craving. The investigators hypothesize that repetitive TMS reduce meth cue craving in meth dependent population compared with sham rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Be volunteers who are dependent on meth and not currently seeking treatment. They must not have received substance abuse treatment within the previous 30 days.
2. Be male or female of any race or ethnic group, between the ages of 18 and 50 years.
3. Meet DSM IV criteria for meth dependence as determined by the MINI International Neuropsychiatric Interview (MINI).
4. Currently be using meth by smoked, oral, or intravenous routes of administration, used meth for a minimum of 2 years and a minimum of an average of 3 times a week in the 30 days prior to screening.
5. Be in stable mental and physical health.
6. If female, test non-pregnant and use adequate birth control. All female subjects will have urine pregnancy tests in all three phases of the study.
7. Be capable of providing written informed consent to participate in this study.
8. Be able to comply with protocol requirements and be likely to complete all study procedures.
9. Live within a 50 mile radius of our research program, have reliable transportation, and have a stable residence for at least the 30 days prior to starting the study.
10. Be willing to abstain from alcohol, marijuana and CNS acting prescription and OTC medications for the 2 week screening and hospitalization phases.
11. Have a positive urine for meth within 72 hours of admission to the hospital phase of the study and have at least one other positive urine for meth during the screening phase.
12. Be right-handed.

Exclusion Criteria:

1. Have current dependence, defined by DSM IV criteria, on any psychoactive substances other than meth, nicotine, or caffeine.
2. Have a history and/or test positive for significant hepatic, renal, endocrine, cardiac, or inflammatory diseases, as well as stroke, seizures, migraine, serious head trauma, or other neurological disorders that might interfere with stability during the study or the acquisition of accurate fMRI scans.
3. If female, have intentions to become pregnant during the study.
4. Have been required by the courts to obtain treatment for meth or some other substance dependence.
5. Be seeking treatment for meth or other substance dependence.
6. Have a medical history or condition considered by the investigators to place the subject at increased risk (implanted ferrous materials or devices) or to decrease the likelihood of study completion.
7. Be anticipating elective surgery or hospitalization within 8 weeks of signing the informed consent agreement.
8. Be on medications in the last 30 days that may alter CNS function or alter fMRI results. Examples of such medications include but are not limited to the following: psychotropics, CNS active anti-hypertensives, steroids, anticonvulsants, antihistamines and CNS OTCs.
9. Have a life time history of major Axis I disorders such as: BPAD, Schizophrenia, PTSD, or Dementia, or have a current history of Major Depression or suicide attempt within 12 months
10. Have a self report of >21 standard alcohol drinks per week in any week in the 30 days prior to screening or a Carbohydrate Deficient Transferrin >3.0%.
11. Be unwilling to use a patch and cease smoking cigarettes for the eight days in the hospital.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Barr MS, Farzan F, Wing VC, George TP, Fitzgerald PB, Daskalakis ZJ. Repetitive transcranial magnetic stimulation and drug addiction. Int Rev Psychiatry. 2011 Oct;23(5):454-66. doi: 10.3109/09540261.2011.618827. PMID 22200135
- [Background] Feil J, Zangen A. Brain stimulation in the study and treatment of addiction. Neurosci Biobehav Rev. 2010 Mar;34(4):559-74. doi: 10.1016/j.neubiorev.2009.11.006. Epub 2009 Nov 13. PMID 19914283
- [Derived] Li X, Malcolm RJ, Huebner K, Hanlon CA, Taylor JJ, Brady KT, George MS, See RE. Low frequency repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex transiently increases cue-induced craving for methamphetamine: a preliminary study. Drug Alcohol Depend. 2013 Dec 1;133(2):641-6. doi: 10.1016/j.drugalcdep.2013.08.012. Epub 2013 Aug 26. PMID 24028801

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Magnetic Stimulation: Transcranial magnetic stimulation (TMS) is a noninvasive brain stimulation technology that can focally stimulate the brain of an awake individual. The brain stimulation techniques could theoretically improve the efficacy of smoking cessation.
  Transcranial Magnetic Stimulation: Active TMS:1 Hz, 100% motor threshold TMS for 15 minutes, total 900 pulses.
  Electrical stimulation instead.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.6) | 32.5 (14.4) | 33.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cue Craving Rating
Description: The subject is asked to rate craving with 0 mm being " no craving at all" and 100 mm representing "the most craving I have ever had".
Time Frame: Change from Baseline in Craving rating 10 minutes after TMS
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 8
scores on a scale | 9.36 (0.75) | 7.92 (0.85)

2. Secondary Outcome: Change in Baseline of Resting Motor Threshold
Description: Resting motor threshold (RMT); on a scale of 0-100 with 100 being most power given to enact a motor response
Time Frame: Baseline to 10 minutes after TMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 8
units on a scale | 47.3 (16.2) | 47.2 (13.5)

3. Secondary Outcome: Change in Cortical Silent Period
Description: Cortical Silent Period is measured in seconds
Time Frame: Baseline and 10 minutes after TMS
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 8
seconds | 0.163 (.053) | .139 (.036)

4. Secondary Outcome: Change Recruitment Curve (RC) Slope
Description: Recruitment Curve (RC) Slope, measured at angle of slope
Time Frame: Baseline and 10 minutes after TMS
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 8
ratio | .272 (.196) | .135 (.073)

ADVERSE EVENTS:
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes